CLINICAL TRIAL: NCT01402661
Title: CorEvitas Rheumatoid Arthritis (RA) Drug Safety & Effectiveness Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Collaborators: University of Massachusetts, Worcester (Other); University of Alabama at Birmingham (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-RA-100
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; psoriatic arthritis; disease registry
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis: Pts presenting to enrolling sites across the US are invited to enroll if eligible.

SUMMARY:
This prospective, non-interventional research registry is designed to study the comparative effectiveness and comparative safety of approved treatments for RA in a cohort of patients cared for by rheumatologists across North America. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
The primary objective for this registry is to systematically collect and document use patterns, effectiveness, and safety of DMARDs (Disease Modifying Anti-Rheumatic Drugs), biologic agents, and any other treatments currently used in the management of RA.

The design is a prospective, non-interventional registry for patients with RA under the care of a rheumatologist. Longitudinal data are collected from both patients and their treating rheumatology providers during routine clinical encounters using a structured and standardized data collection method. The scope of data collection includes but is not limited to patient demographics, disease duration, medical history (including all prior and current treatments for RA), smoking status, alcohol use, disease activity and severity, pain, as well as other clinician- and patient-reported outcomes, comorbidities and adverse events, infections, hospitalizations, and other targeted safety outcomes. After the enrollment visit, RA patients and physicians will complete the follow-up questionnaires during regularly scheduled clinical encounters. The goal is to collect data from patients and providers at six month intervals. Adverse events may be volunteered spontaneously by the subject, or be discovered as a result of general questioning by the Investigator. During all CorEvitas related visits with the Investigator, subjects will be questioned regarding the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age or older.
2. Be able and willing to provide written consent for participation in the registry as well as Personally Identifiable Information (PII) that includes Full Name and Date of Birth at a minimum.
3. Have been diagnosed with rheumatoid arthritis by a rheumatologist.
4. Meet at least one of the following criteria:

(A) Currently receiving an Eligible Medication** that was started within 365 days of the Enrollment Visit.

i. A temporary interruption of an Eligible Medication is allowed if the interruption in treatment lasted <180 days.

(B) Prescribed or receiving the first dose of an Eligible Medication** on the day of the Enrollment Visit.

(C) Diagnosed with RA within 365 days of the Enrollment Visit regardless of treatment regimen ("Early RA").

Exclusion Criteria:

The patient must not:

1. Have a diagnosis of Juvenile idiopathic arthritis (JIA), Psoriatic arthritis (PsA), Spondyloarthritis (SpA), Ankylosing spondylitis (AS), Systemic lupus erythematosus (SLE), or any other form of autoimmune inflammatory arthritis.
2. Be starting only a non-eligible medication, unless the patient was diagnosed with RA within 365 days of the Enrollment Visit. Non-eligible medications include conventional DMARDs - for example methotrexate, sulfasalazine, leflunomide, etc. - and including prednisone.
3. Be participating in or planning to participate in a double-blind randomized clinical trial of an RA drug. Of note, concurrent participation in another observational registry or open-label Phase 3b/4 trial is not excluded.

   Early Follow-Up Visit Criteria

   To be eligible for an early CorEvitas Follow-Up Visit that is conducted <150 days since the last registry visit, the following conditions must be met:
4. A follow-up set of questionnaires should always be completed whenever a registry subject is being prescribed or receiving the first dose of a new (different) Eligible Medication** at a routine office visit. If this occurs less than 150 days from the previous visit at which CorEvitas questionnaires had been completed, it is considered an "Early Follow-Up Visit." The next anticipated visit that follow-up questionnaires would be completed would be calculated off the Early Follow-up Visit date (=>150 days). Prior use of an Eligible Medication** does not exclude a patient from an Early Follow-Up visit.

   * Eligible Medications are biologics, biosimilars, and JAK-inhibitors FDA-approved for the treatment of RA. Prior use of an Eligible Medication does not exclude a patient from enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the CorEvitas Data Collection Program during regularly-scheduled office visits. Selected rheumatologists are invited to participate as investigators in the CorEvitas Data Collection Program. Physicians are selected carefully in an effort to ensure enrollment of subjects that represent a reasonable representation of a cross-section of the population throughout the country with rheumatic diseases. All potential sites are screened for clinical research experience and adherence to GCP (Good Clinical Practice) guidelines
Sampling Method: Non-Probability Sample
Enrollment: 91758 (Estimated)
Dates: Start 2002-02 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Patterns, effectiveness, and safety of DMARDs, biologic agents and any other treatments currently used in the management of RA | Data are collected on subjects for as long as they consent to remain in the study

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kremer, MD, Study Director — Center for Rheumatology
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litman HJ, Sheffield KM, Pugach O, Shan M, Lakin P, Cui ZL, Curtis SE, Johnston JA, Harrold LR. Applying Bias Correction Methods to Build Hybrid Controls Using Real-World Patients for a Phase IIb Randomized Controlled Trial of Baricitinib for Rheumatoid Arthritis. Pharm Stat. 2025 Jul-Aug;24(4):e70020. doi: 10.1002/pst.70020. PMID 40493525
- [Derived] Harrold LR, Bingham CO, Pope JE, O'Brien J, Moore PC, Roberts-Toler C, Yu M, Sweet LL, Shelbaya A, Masri KR. Effectiveness of tofacitinib versus tumor necrosis factor inhibitors and in those receiving tofacitinib as different lines of therapy in patients with rheumatoid arthritis: results from the United States CorEvitas Rheumatoid Arthritis Registry. Clin Rheumatol. 2025 Feb;44(2):635-648. doi: 10.1007/s10067-024-07245-3. Epub 2024 Dec 20. PMID 39707042
- [Derived] Pappas DA, Blachley T, Best JH, Zlotnick S, Reiss WG, Emeanuru K, Kremer JM. Durability of Response to Tocilizumab Therapy in Rheumatoid Arthritis: Data from the US-Based Corrona Rheumatoid Arthritis Registry. Rheumatol Ther. 2021 Mar;8(1):467-481. doi: 10.1007/s40744-021-00285-0. Epub 2021 Feb 25. PMID 33630272
- [Derived] Pappas DA, Blachley T, Zlotnick S, Best J, Emeanuru K, Kremer JM. Methotrexate Discontinuation and Dose Decreases After Therapy With Tocilizumab: Results From the Corrona Rheumatoid Arthritis Registry. Rheumatol Ther. 2020 Jun;7(2):357-369. doi: 10.1007/s40744-020-00200-z. Epub 2020 Mar 30. PMID 32232740
- [Derived] Pappas DA, Etzel CJ, Zlotnick S, Best J, Blachley T, Kremer JM. Patterns of Prednisone Use in Patients with Rheumatoid Arthritis Initiating Treatment with Tocilizumab in Routine US Clinical Practice. Rheumatol Ther. 2019 Sep;6(3):421-433. doi: 10.1007/s40744-019-0162-6. Epub 2019 Jun 25. PMID 31240499
- [Derived] Mease PJ, Collier DH, Saunders KC, Li G, Kremer JM, Greenberg JD. Comparative effectiveness of biologic monotherapy versus combination therapy for patients with psoriatic arthritis: results from the Corrona registry. RMD Open. 2015 Dec 30;1(1):e000181. doi: 10.1136/rmdopen-2015-000181. eCollection 2015. PMID 26819748
- [Derived] Harrold LR, Reed GW, Magner R, Shewade A, John A, Greenberg JD, Kremer JM. Comparative effectiveness and safety of rituximab versus subsequent anti-tumor necrosis factor therapy in patients with rheumatoid arthritis with prior exposure to anti-tumor necrosis factor therapies in the United States Corrona registry. Arthritis Res Ther. 2015 Sep 18;17(1):256. doi: 10.1186/s13075-015-0776-1. PMID 26382589
- See also: CorEvitas home page: — https://www.corevitas.com/